CLINICAL TRIAL: NCT00133042
Title: The Effect of Omalizumab on Airway Responsiveness to Adenosine in Patients With Poorly Controlled Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CIGE025 US06
Record Dates: First submitted 2005-08-19; First posted 2005-08-22 (Estimated); Last update posted 2011-09-20 (Estimated); Status verified 2009-02

CONDITIONS: Asthma
Keywords: anti-IgE, omalizumab
MeSH Terms: conditions — Asthma | interventions — Omalizumab

INTERVENTIONS:
Drug: omalizumab

SUMMARY:
The purpose of this study is to determine whether the addition of omalizumab in patients with poorly controlled asthma (because of poor adherence) will decrease allergic airway inflammation and improve asthma control.

DETAILED DESCRIPTION:
Patients with moderate to severe allergic asthma who are poorly adherent to inhaled corticosteroids (ICS) have persistent airway inflammation that results in excessive morbidity and sometimes death. Omalizumab (OMB), an anti-IgE monoclonal antibody decreases the release of mediators from mast cells, reduces the frequency of exacerbations and allows a reduction in ICS dose. However, there are no data on the effects of OMB on airway inflammation. Bronchoprovocation with adenosine 5' monophosphate (AMP) is a robust and sensitive non-invasive measure of allergic airway inflammation, but the effect of OMB on this surrogate marker has not been previously reported. Based upon the mechanisms of actions of OMB and AMP and the fact that OMB will be administered at 2-4 week intervals in the clinic (i.e., direct observed therapy), it is our hypothesis that treatment with this new agent will reduce airway responsiveness to AMP and compensate for poor adherence to ICS.

To test this hypothesis, we will select 16 patients (6-26 yrs) with a total IgE of 30-1300 IU/ml, sensitivity to at least one allergen, an FEV1 ≥ 60% predicted, and documented poor adherence to ICS with inadequate asthma control. Subjects will be randomized to receive OMB (150-375 mg subcutaneously) or placebo every 2-4 weeks for four months each, in a double-blind, crossover manner with a 3 month washout period between treatments. Spirometry will be measured before each injection and at the end of each treatment period. The concentration of AMP that will provoke a 20% decrease in FEV1 (PC20 FEV1) and a free IgE serum concentration will be measured before and at the end of each treatment period. After randomization, a 5-day course of oral prednisone will be administered whenever bronchodilator-unresponsive symptoms persist or FEV1 is < 60% predicted. ANOVA for repeated measures will be used to evaluate differences between treatments in Δ PC20 (primary endpoint) and Δ FEV1, while the Friedman Statistic will be used to evaluate differences in the number of short courses of prednisone. The results of this study will provide new information on the extent to which OMB decreases airway responsiveness to AMP (i.e. allergic airway inflammation) and whether this new therapy will fill an unmet need for patients who have inadequately controlled asthma because of poor adherence to inhaled corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking subjects
* 6-26 years of age
* Evidence of poor asthma control
* Adherence to ICS < 50% of doses prescribed over a minimum of 3 months
* Baseline FEV1 > 60% of predicted
* PC20 AMP < 60 mg/ml
* Able to perform American Thoracic Society (ATS)-acceptable and reproducible spirometry

Exclusion Criteria:

* Cigarette smoking/use of marijuana
* Pregnancy
* Respiratory infections in past six weeks
* History of acute allergic reaction to asthma/allergy medication
* Total dose requirement of omalizumab more than 375 mg every two weeks
* Inability to withhold required medications before challenge
* Abnormal electrocardiogram (ECG)

Ages: 6 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16
Dates: Start 2004-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
adenosine, PC20, forced expiratory volume in one second (FEV1)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Hendeles, PharmD, Principal Investigator — University of Florida
Locations (1):
- University of Florida Asthma Research Lab, Gainesville, Florida, United States

REFERENCES:
- [Derived] Hendeles L, Khan YR, Shuster JJ, Chesrown SE, Abu-Hasan M. Omalizumab therapy for asthma patients with poor adherence to inhaled corticosteroid therapy. Ann Allergy Asthma Immunol. 2015 Jan;114(1):58-62.e2. doi: 10.1016/j.anai.2014.10.012. PMID 25528738